CLINICAL TRIAL: NCT07014683
Title: INtegral Cognitive REMediation for Depression (INCREM). Multicentric Randomized Clinical Trial to Investigate Feasibility and Efficacy (Phase II)
Brief Title: Integral Cognitive Remediation for Depression
Acronym: INCREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-RID-2021-07
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: cognitive symptoms; cognitive remediation; rehabilitation; functional recovery; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Neurobehavioral Manifestations | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INCREM (Experimental): 12-session integral cognitive remediation program specifically designed for depression.
  Interventions: Behavioral: INCREM
- Psychoeducation (Active Comparator): 12-session psychoeducation program for depression
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: INCREM — This is a specifically designed program to improve psychosocial functioning which targets cognitive symptoms.
  Other Names: cognitive remediation
  Arms: INCREM
Behavioral: Psychoeducation — This is a 12-session psychoeducation program designed as an active comparator for the current trial
  Arms: Psychoeducation

SUMMARY:
The goal of this clinical trial is to learn if INCREM intervention can improve psychosocial functioning in patients with remitted major depressive disorder. The main question it aims to answer are:

Does INCREM improve psychosocial functioning compared to psychoeducation? Does the benefits of INCREM remain after six months of the intervention compared to psychoeducation?

Researchers will compare two arms: INCREM; psychoeducation to see if psychosocial functioning improves.

Participants will be allocated to:

* INCREM
* Psychoeducation
* TAU.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 y.o. and beyond with a remitted or active episode of major depression (DSM-5 criteria; maximum score of 18-20 on the HDRS-17) showing cognitive symptoms (scores below 80 on the SCIP) with functional difficulties (scores above 12 on the FAST).

Exclusion Criteria:

* IQ below 85;
* any unstable or inadequately-treated medical condition that may affect neuropsychological performance;
* being under drug treatment in the last 4 weeks with glucocorticoids, probiotics, non-steroidal anti-inflammatory drugs, bile acid sequestrants, immunosuppressive drugs, anti-histamines, mast cell stabilizers, and antioxidant supplements;
* use of systemic antibiotics the last 2 months;
* presence of any comorbid psychiatric condition, other than personality disorders or nicotine use disorders, in the last three months;
* accomplish criteria for severe treatment resistant depression;
* patients who had received electroconvulsive therapy in the previous year;
* patients receiving any other structured psychological intervention in the 3 months prior to the study;
* not having the necessary electronic means (computer or tablet) or internet connection to be able to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2023-08-13 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Functioning Assessment Short Test (FAST) | From enrollment to the end of treatment (12 weeks) and to the end of follow-up (6 months)
  The FAST is a valid, widely used instrument to test psychosocial functioning. The main outcome measure will be the percentage of change in FAST scores between T0 and T1 and T2.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17 items (HDRS_17) | From enrollment to the end of treatment (12 weeks) and to the end of follow-up (6 months)
  This scale is used to rate the severity of depression symptoms by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms.
Screening for Cognitive Impairment in Psychiatry (SCIP) | From enrollment to the end of the intervention (12 weeks) and to the end of the follow-up (6 months)
  The SCIP is a brief and easy-to-administer tool, requiring the test sheet, a clock and a pencil only, specifically targeting psychiatric populations.
Perceived Deficits Questionnaire for Depression (PDQ-R) | From enrollment to the end of the intervention (12 weeks) and to the end of follow-up (6 months)
  The PDQ-D is a self-reported scale for monitoring cognitive dysfunction in patients with major depression. The PDQ-D is a modified version of the original PDQ, which was developed to assess cognitive symptoms in patients with multiple sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Portella, Dr, Principal Investigator — Fundació Institut de Recerca Hospital de la Santa Creu i Sant Pau
Locations (1):
- Institut de Recerca Sant Pau- Mental Health Group, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided